CLINICAL TRIAL: NCT02217995
Title: A Pilot Randomized Trial Testing Mindfulness-Based Cognitive Therapy in a Clinical Sample of OCD Patients
Brief Title: Mindfulness-Based Cognitive Therapy in a Clinical Sample of OCD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Neil Rector, Research Scientist and Psychologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 138-2014
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Mindfulness-Based Cognitive Therapy; Mindfulness
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness-Based Cognitive Therapy (MBCT) (Experimental): MBCT will be delivered in ten 2.5 hour group sessions with 15 participants per group.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy (MBCT)
- Waitlist (No Intervention): Wait list as per usual.

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy (MBCT) — MBCT teaches patients to become more aware of, and to relate differently to, their thoughts, feelings, and bodily sensations. Through MBCT, patients will learn skills that allow them to disengage from habitual ("automatic") dysfunctional cognitive routines, such as obsessional thinking. As an example, patients are encouraged to relate to thoughts and feelings as passing events in the mind, rather than to identify with them or treat them as accurate representations of reality. The MBCT protocol for OCD patients is adapted from Segal et al.'s original MBCT manual for depression (Segal, Williams & Teasdale, 2002).
  Arms: Mindfulness-Based Cognitive Therapy (MBCT)

SUMMARY:
Obsessive Compulsive Disorder (OCD) is a chronic and debilitating disorder known to have reported lifetime prevalence in the range of 2%. OCD is most commonly treated with Cognitive Behavioural Therapy (CBT) and/or pharmacotherapy. However, some studies suggest challenges with CBT in retaining gains long term, and while 60-80% of OCD patients respond to SRI treatment, partial symptom reduction is substantial. Investigations into the effectiveness of alternative, cost-effective treatment modalities are thus needed. Mindfulness, defined as paying attention in a particular way (on purpose, in the present moment and nonjudgmentally), promotes awareness and attention to internal experience and has been shown to reduce symptoms of anxiety and depression. A number of controlled studies have found Mindfulness-Based Cognitive Therapy (MBCT) to be effective for depression, social anxiety disorder, and generalized anxiety disorder, but few have tested its effect on obsessive compulsive disorder (OCD). Moreover, those studies examining MBCT in OCD focused on clinical case studies and non-clinical samples. This study proposes to examine the effect of MBCT in clinical practice, in a randomized sample of patients with OCD whom are on a clinic wait list. As patients are allocated to the wait list, they will be randomly assigned to receive either 10 weeks of group MBCT or wait list as per usual. It is hypothesized that subjects randomly assigned to the MBCT treatment group, compared to those in the wait list control group, will see greater reductions in self-reported measures of OCD symptom severity and improvement in other measures of mindfulness, mood and level of functioning. The results of this pilot study, if successful, will provide evidence towards another route by which patients can improve their OCD while waiting for clinic services or consultation. Results will also lend more evidence as to whether MBCT is effective as a stand-alone treatment for clinical OCD, which will inform further investigations into the potential addition of mindfulness techniques to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Referred for treatment services at the Frederick W. Thompson Anxiety Disorder Centre at Sunnybrook Health Sciences Centre
* Primary Diagnosis of OCD
* Ability to communicate in written and spoken English

Exclusion Criteria:

* Those with active substance abuse/dependence within 3 months
* Suspected organic pathology
* Recent suicide attempt/active suicidality
* Current self-injurious behaviour
* Active bipolar or psychotic disorder
* Previous completion of an MBCT course (≥ 8 weeks)
* Previous completion of an OCD-specific course of CBT (≥ 8 weeks)
* Previous completion of a general course of CBT (≥ 8 weeks) in the past 3 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-09; Primary Completion 2017-08 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Change in Symptom Severity from Baseline in OCD Measures | 10 weeks
  OCD measures will include: a self-report version of the Yale-Brown Obsessive Compulsive Scale (YBOCS-SR), the Obsessive Compulsive Inventory -Revised (OCI-R), consisting of six subscales (Washing, Checking, Ordering, Obsessing, Hoarding and Neutralising), and the Obsessive Beliefs Questionnaire-44 (OBQ-44), a measure of three OCD-related belief domains (Perfectionism/Certainty, Importance/Control of thoughts, and Responsibility/Threat estimation)

SECONDARY OUTCOMES:
Change in Level of Impairment from Baseline | 10 weeks
  The Sheehan Disability Scale will be used to measure level of functional impairment in three inter-related domains (work/school, social and family life).
Change in Mood from Baseline | 10 weeks
  The Beck Depression Inventory -II (BDI-II), will be used to assess depression severity.
Change in Mindfulness from Baseline | 10 weeks
  Mindfulness measures include: The Five Facet Mindfulness Questionnaire (FFMQ), used to measure the five constructs central to mindfulness (Observing, Describing, Acting with Awareness, Non-judgment of Inner Experience, and Non-reactivity to Inner Experience), and the the Self-Compassion Scale-Short Form (SCS-SF) measuring 6 components of self-compassion (Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness & Over-Identification).
Retention of Gains at Follow-up | 16 weeks
  All self-report measures will be re-administered at 6-week follow-up to measure robustness of gains post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Frederick W. Thompson Anxiety Disorders Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada